CLINICAL TRIAL: NCT02429635
Title: Workplace Health and Wellness Promotion: Investigating the Effects of a Team-based Intervention on Individual Motivation and Enhanced Physical Activity, Health and Work-functioning
Brief Title: My Exercise. A Team-based Workplace Intervention for Increased Exercise
Acronym: Myexercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Hallgeir Halvari, Professor II, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013/294; 227874 (Other Grant/Funding Number: The Research Counsil of Norway)
Record Dates: First submitted 2015-04-14; First posted 2015-04-29 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Inactivity/Low Levels of Exercise
Keywords: Exercise; lifestyle diseases; well-being
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- My exercise (Experimental): Health Screening I and II Questionnaires on health and lifestyle, physiological test of fitness, physiological health tests and blood profile - compiled in a health profile report. Individual guidance and advice from professional health advisor.
  Team-workshop I and II A 2 hours' workshop lead and facilitated by a trained and professional health advisor. It consists of short talks on exercise and health, and on health behavior change and motivation in addition to work with self-reflection and discussion tasks. Competence, support and advice during 2. workshp.
  Exercise groups Small groups with similar exercise level and ambitions who support each other in their efforts to establish new exercise habits according to their individual exercise plan.
  Interventions: Behavioral: My exercise
- Control group - delayed intervention (Experimental): Health Screening I and II Questionnaires on health and lifestyle, physiological test of fitness, physiological health tests and blood profile - compiled in a health profile report. Individual guidance and advice from professional health advisor.
  Team workshops and training groups The control groups will consist of teams that will receive the team-based health promotion measures about 9 months after the Team-based health promotion measures group.
  Interventions: Behavioral: My exercise

INTERVENTIONS:
Behavioral: My exercise — Health Screening I and II Questionnaires on health and lifestyle, physiological test of fitness, physiological health tests and blood profile - compiled in a health profile report. Individual guidance and advice from professional health advisor.
  Team-workshop I and II A 2 hours' workshop lead and facilitated by a trained and professional health advisor. It consists of short talks on exercise and health, and on health behavior change and motivation in addition to work with self-reflection and discussion tasks. Competence, support and advice during 2. workshop.
  Exercise groups Small groups with similar exercise level and ambitions who support each other in their efforts to establish new exercise habits according to their individual exercise plan
  Other Names: A team-based health promotion intervention

SUMMARY:
The aim of this research study is to assess the effectiveness of an intervention on exercise and health, and to contribute to the understanding of how team-based worksite health promotion programs should be designed in order to increase and maintain exercise among employees. The study design is a randomized controlled trial.

There are a number of different theories on the subject of how to affect motivation for health behavior change. This study is based on the tenets of Self-Determination Theory (SDT) in combination with elements from Motivational Interviewing and in accordance with the Health Promotion Guidelines developed by the National Institute of Health and Clinical Excellence, NICE.

It is assumed that if such a program is designed and offered in a manner that satisfies the participants' sense of autonomy, competence and relatedness, this will affect the quality of the participants' self-regulated motivation and perceived competence for exercise and lifestyle changes. As a consequence, a large proportion of the participants will adhere to the program and increase their exercise both in the short (5 months) and long term (8 months).

The following research questions will be:

1. Would a team-based health and exercise promotion intervention designed to be needs supportive, relative to a control group:

   1. Influence increases in exercise levels, improved aerobic fitness, reduced blood pressure, and decreases in waist circumference, and Body mass index (BMI), in addition to changes in body composition in terms of reduced percentage of fat and increased percentage of muscles?
   2. Influence increases in psychological well-being?
   3. Influence increases in perceived investment in employees' health competence, which would positively predict affective organizational commitment and job performance, and negatively predict turnover intentions?
   4. Influence decreases in sickness absenteeism?
2. If so, would changes in psychological needs support, autonomous motivation for exercise, perceived competence and self-efficacy in exercise mediate these effects?

DETAILED DESCRIPTION:
The principal contribution of this study is the understanding of whether and how a SDT-based intervention affects the participants' degree of autonomous motivation and perceived competence for exercise, and as a consequence behavioral change in the form of increased and regular exercise. That is, the psycho-social processes which are unfolding during the intervention, and caused by the intervention.

The intervention is implemented in a worksite setting and connected to a team-based health promotion program.

This is a cluster-randomized two-group trial that compares a group-based intervention with a control group. Cluster-randomization will be carried out at the level of physical location consisting of two work teams each.

Pre- and post-test assessments will be carried out during an individual health screening consisting of physiological tests and cross-sectional data collection in the form of quantitative and standardized questionnaires. The results are compiled in a health profile report. Participants are offered a 15-20 minutes individual consultation with the professional health advisor in order to explain the findings, answer quesdtions and giving healht recommendations.

A small collection of the questionnaires and some qualitative interviews will be applied in order to collect data on relevant variables during the intervention period as well as to assess fidelity and participants' perceptions of the intervention.

The intervention consists of three elements; two team-workshops, exercise support group meetings and a workbook for self-reflection and planning. The intervention will be carried out by two health advisors professionals (physiotherapist) trained in order to facilitate and lead the team-workshops in a need supportive manner.

ELIGIBILITY:
Inclusion Criteria:

* Employment at the Norwegian Post
* Position of 40% or more

Exclusion Criteria:

* Temporary employment that lasts for less than 12 months

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Changes from baseline levels of regular exercise (International Physical Activity Index (IPAI) | T1: baseline, T2: post-test 5 months, T3: post-test 8 months
  Assessed by a self reported questionnaire: International Physical Activity Index (IPAI). (Kurtze et al., 2008)
Changes from baseline cardiovascular endurance/aerobic fitness (Astrand-Rhyming Cycle Ergometer Test) | T1: baseline, T2: Post-test 5 months
  Assessed by Astrand-Rhyming Cycle Ergometer Test. This ia submaximal cycle ergometer aerobic fitness test (Astrand, 1960).

SECONDARY OUTCOMES:
Changes from baseline Systolic Blood Pressure (measured manually by means of an auscultatory technique with a mercury column or mechanical aneroid sphygmomanometer) | T1: baseline, T2: Post-test 5 months
  Changes will be measured manually by means of an auscultatory technique with a mercury column or mechanical aneroid sphygmomanometer.
Changes from baseline body weight and composition (Tanita Scale) | T1: baseline, T2: post-test 5 months
  Tanita Scale - Body Composition Tracking Charts, Body Mass Index (BMI) (Keys et al., 1972), and waist circumference
Changes from baseline self-regulated motivation for exercise (Behavioral Regulation in Exercise Questionnaire (BREQ-2) | T1: Prbaseline, T2: post-test 5 months, T3: post-test 8 months
  Assessed by a self-reporting questionnaire Behavioral Regulation in Exercise Questionnaire (BREQ-2), Mullan et al.(1997)
Changes from baseline basic psychological needs satisfaction in exercise (Basic Psychological Needs in Exercise Scale (BPNES) | T1: baseline, T2: post-test 5 months, T3: post-test 8 months
  Assessed by self-reporting questionnaire:The Basic Psychological Needs in Exercise Scale (BPNES) Vlachopoulos and Michailidou (2006)
Changes from baseline perceived self-efficacy in exercise (Self-efficacy in Exercise Scale) | T1: baseline, T2: post-test 5 months, T3: post-test 8 months
  Assessed by self-reporting questionnaire: Self-efficacy in Exercise Scale, Fuchs and Schwarzer (1994)
Changes from baseline perceived competence for exercise (Perceived Competence for Exercise Scale) | T1: baseline, T2: post-test 5 months, T3: post-test 8 months
  Assessed by self-reporting questionnaire: Perceived Competence for Exercise Scale, Williams and Deci (1996)
Changes from baseline perceived work effort and work performance (Effort and Quality of Work) | T1: baseline, T2: post-test 5 months, T3: post-test 8 months
  Assessed by self-reporting questionnaire: Effort and Quality of Work, Kuvaas(2006)
Changes from baseline turnover intentions (Current Turnover Intentions) | T1: baseline, T2: post-test 5 months, T3: post-test 8 months
  Assessed by two self-reporting questionnaires: Current Turnover Intentions(O'Driscoll and Beehr, 1994) and Past Year Turnover Intentions (Luchak and Gellatly, 2007)
Changes from baseline attitutes towards work and employer, affective commitment (Organizational Commitment, Affective Commitment Sub-scale) | T1: baseline, T2: post-test 5 months, T3: post-test 8 months
  Assessed by self-reporting questionnaire Organizational Commitment, Affective Commitment Sub-scale, Allen and Meyer (1990)
Changes from baseline perceived investment in health competence by employer (Perceived investment in employee development (PIED) adjusted to health competence) | T1: baseline, T2: post-test 5 months, T3: post-test 8 months
  Assessed by self-reporting questionnaire: Perceived investment in employee development (PIED) adjusted to health competence, Kuvaas and Dysvik (2009)
Changes from baseline satisfaction with life and well-being in general (Satisfaction in Life Scale, and Subjective Vitality) | T1: baseline, T2: post-test 5 months, T3: post-test 8 months
  Assessed by two self-reporting questionnaires: Satisfaction in Life Scale, Pavot and Diener (1993), and Subjective Vitality, Ryan and Frederick (1997)
Changes from baseline positive and negative affect (Positive and Negative Affect Scale (PANAS) | T1: baseline, T2: post-test 5 months, T3: post-test 8 months
  Assessed by self-reporting questionnaire: Positive and Negative Affect Scale (PANAS) Watson et al. (1988)
Changes from baseline somatic symptoms burden (Somatic Symptom Scale (SSS-8) | T1: baseline, T2: post-test 5 months, T3: post-test 8 months
  Assessed by self-reporting questionnaire: The Somatic Symptom Scale (SSS-8), Gierk et al. (2014)
Changes from baseline sickness absence and presenteeism | T1: baseline, T2: post-test 5 months, T3: post-test 8 months
  Assesses by self-reporting questionnaire: Sickness absence and presenteeism, Aronsson and Lindh (2004)
Changes from baseline perceived support from work peers related to exercise (The Health Care Climate Questionnaire (HCCQ) | T1: baseline, T2: post-test 5 months, T3: post-test 8 months
  Assessed by self-reporting questionnaire: The Health Care Climate Questionnaire (HCCQ), Williams et al., 1996
Changes from baseline perceived support form work peers related to exercise (The Health Care Climate Questionnaire (HCCQ) adjusted to work peers) | T1: baseline, T2: post-test 5 months
  Assessed by self-reporting questionnaire: The Health Care Climate Questionnaire (HCCQ) adjusted to work peers, Williams et al., 1996.
Changes from baseline sickness absence | T1: baseline, T2: post-test 5 months
  Assessed by self-reporting questionnaire: Sickness absence and presenteeism, Aronsson and Lindh, 2004.

CONTACTS AND LOCATIONS:
Overall Officials: Hallgeir Halvari, Professor, Study Chair — Norwegian School of Sport Sciences
Locations (1):
- Norwegian School of Sport Science, Oslo, Norway

REFERENCES:
- [Derived] Pedersen C, Halvari H, Olafsen AH. Worksite physical activity intervention and somatic symptoms burden: The role of coworker support for basic psychological needs and autonomous motivation. J Occup Health Psychol. 2019 Feb;24(1):55-65. doi: 10.1037/ocp0000131. Epub 2018 Aug 16. PMID 30113178